CLINICAL TRIAL: NCT01740076
Title: Effect of Soy Nuts on Blood Pressure, Lipids and Inflammation in Postmenopausal Women
Brief Title: Soy Nuts and Cardiovascular Risk in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2001P001604
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Postmenopausal Women
Keywords: isoflavones, hypertension, soy, diet, nutrition, women, inflammation, hot flashes
MeSH Terms: conditions — Hypertension; Inflammation; Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- soy nuts (Experimental): 25 g of soy nuts provided daily to the subjects and they were counseled to replace 25 g of protein in their therapeutic lifestyle change (TLC) diet with the soy. TLC diet consisted of 30% of energy from total fat (<7% saturated fat, 12% monounsaturated fat and 11% polyunsaturated fat), 15% from protein and 55% from carbohydrate; less than 200 mg of cholesterol per day and 1200 mg of calcium and 2 fatty fish meals per week. Those ingesting suboptimal dietary calcium were given calcium carbonate supplementation.
  Interventions: Other: soy nuts
- Therapeutic lifestyle change diet (Other): Counseling on therapeutic lifestyle change diet consisting of 30% of energy from total fat (<7% saturated fat, 12% monounsaturated fat and 11% polyunsaturated fat), 15% from protein and 55% from carbohydrate; less than 200 mg of cholesterol per day and 1200 mg of calcium and 2 fatty fish meals per week. Those ingesting suboptimal dietary calcium were given calcium carbonate supplementation.
  Interventions: Other: soy nuts

INTERVENTIONS:
Other: soy nuts

SUMMARY:
To determine the effect of a whole soy food, dietary soy nuts, on blood pressure, lipid levels, inflammation and menopausal symptoms in postmenopausal women.

DETAILED DESCRIPTION:
The present study examines the effect of a whole soy food, soy nuts (dry roasted soybeans), added to the Therapeutic Lifestyle Change diet on blood pressure, lipids, inflammation and menopausal symptoms in postmenopausal hypertensive and normotensive women in a randomized crossover trial during an 8-week period. We sought to determine whether dietary soy had an additional benefit to the currently recommended heart healthy diet.

ELIGIBILITY:
Inclusion Criteria:

* Women with absence of menses for at least 12 months or irregular periods and hot flashes.

Exclusion Criteria:

* were current cigarette smoking or smoking in the previous year;
* clinical coronary artery disease, peripheral artery disease, or cerebrovascular disease;
* known diabetes mellitus or a fasting glucose level of 126 mg/dL or greater;
* a history of breast cancer; a fasting triglyceride level greater than 400 mg/dL; systolic BP of 165 mm Hg or greater or diastolic BP of 100 mm Hg or greater;
* untreated hypothyroidism; systemic or endocrine disease known to affect lipid, mineral, or bone metabolism;
* and consumption of more than 21 alcoholic drinks per week.
* Use of lipid-lowering drugs, hormone therapy, medications for osteoporosis, and soy products was discontinued for 2 months before entering the study. Participants took a multivitamin but no additional vitamin or mineral supplements or other soy products during the study.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2001-09; Primary Completion 2004-07 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks
  stratified by hypertensive status (normal BP, prehypertension, hypertension)

SECONDARY OUTCOMES:
lipid levels | 8 weeks
  stratified by hypertension status (normotensive or hypertensive)
inflammatory markers | 8 weeks
  stratified by hypertensive status (normotensive or hypertensive)
menopausal symptoms | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francine Welty, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Acharjee S, Zhou JR, Elajami TK, Welty FK. Effect of soy nuts and equol status on blood pressure, lipids and inflammation in postmenopausal women stratified by metabolic syndrome status. Metabolism. 2015 Feb;64(2):236-43. doi: 10.1016/j.metabol.2014.09.005. Epub 2014 Oct 5. PMID 25441251